CLINICAL TRIAL: NCT01675245
Title: Velcade (Bortezomib for Injection) Observational Study
Brief Title: An Observational Study of Chinese Multiple Myeloma Patients Treated With Velcade
Status: Completed | Type: Observational
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR006373; 26866138MMY4031 (Other: Xian-Janssen Pharmaceutical Ltd., China); VEL-CHN-MA-01 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Cancer; Velcade; Bortezomib; Chinese patients
MeSH Terms: conditions — Multiple Myeloma; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Velcade: Velcade, 1.3 mg/m2/dose, administered intravenously on days 1, 4, 8 and 11, for 2 weeks.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Velcade will be administered as per the recommended regimen. (Velcade, 1.3 mg/m2/dose, administered intravenously on days 1, 4, 8 and 11, for 2 weeks)

SUMMARY:
The purpose of this study is to acquire information on the usage, effectiveness, safety, and levels of health care resource utilization associated with Velcade therapy in recurrent and refractory multiple myeloma patients who are initiating Velcade and various combination therapies within the approved indication in a naturalistic setting.

DETAILED DESCRIPTION:
This is a national, multi-center (study conducted in multiple sites), non-interventional (a scientific study where one or more investigators monitor one or more patients being treated with the same medication), observational study (a scientific study to make a clear and easy understanding of the cause and effect relationship) of Chinese Multiple Myeloma patients treated with Velcade. The study consists of 3 phases, including, screening phase, treatment phase, and follow up phase. In the screening phase, data will be collected on the basis of patient's demographic status, components of disease severity assessment, and potential prognostic factors. Data on prior cancer treatments will be collected retrospectively at baseline for patients receiving cancer treatment prior to receiving Velcade. In the treatment phase, Velcade is administered intravenously for a 2-week treatment period followed by a 10-day rest period. Each treatment cycle consists of 21 days. Prospective (in which the participants are first identified and then followed forward as time passes) observational data will be collected during treatment with Velcade. In the follow up phase, patients will be followed for up to three years to document long-term survival data. For patients who reinitiate Velcade, data collection should follow Velcade treatment period documentation process. Safety evaluations will be based on the incidence, intensity, and types of adverse events. The total duration of the study is set prospectively for three years from the date of the patients' initiation of Velcade.

ELIGIBILITY:
Inclusion Criteria:

* Must give informed consent in agreement with local legislation
* Must not have any contraindication listed in package insert

Exclusion Criteria:

* Patients currently participating in another investigational study of Velcade or any other medication
* Patients with severe hepatic or renal impairment
* Patients with platelet count below 25000/μl
* Patients who are considered disqualified for the study by the investigators

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with multiple myeloma (based on standard diagnosis criteria), initiating Velcade therapy within the approved indication.
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2006-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Information on treatment sequence for Velcade therapy | Baseline (Day -1) to Day 21
  Treatment sequence or the line of therapy will be considered on Velcade utilization.
Information on dosage of Velcade | Baseline to Day 21
  Dosage of Velcade will be considered on Velcade utilization. The unit of dosage will be milligram per square meter body surface area.
Information on duration of Velcade therapy | Baseline to Day 21
  Duration of Velcade therapy will be measured on Velcade utilization. The unit of duration will be number of days or the length of the course of therapy.
Information on patient diagnosis for Velcade therapy | Baseline to Day 21
  Diagnosis of patients will be considered on Velcade utilization.
Number of patients with disease response or progression | Up to 3 years
  Complete response (CR), near complete response (complete response with positive immunofixation; nCR), partial response (PR), minimal response (MR), stable disease (SD), progressive disease (PD), or relapse from CR (RCR); the methods and criteria used to evaluate the responses will be chosen by the physician and recorded.
Time to response | Up to 3 years
  Time to response is calculated from the start date of the cycle of Velcade therapy.
Duration of response | Up to 3 years
  Duration of response is calculated from the date on which response is documented until PD, RCR, death, or study termination occurs.
Time to progression | Up to 3 years
  Time to progression is calculated from the date on which response is documented until PD or RCR occurs.
Survival status | Up to 3 years
  Survival status is calculated from the start of Velcade therapy until death; to be monitored, to the extent possible, beyond the end of Velcade therapy, up to the end of the study period.
Number of patients with adverse events | Up to 3 years
  Safety criteria will be considered for new skeletal events (fractures, radiotherapy of bone, operation on the bone, spinal cord compression), infection and haematological toxicity (with greater than or equal to grade 3 using WHO Common Toxicity Criteria [WHO CTC]), and any neurotoxic events by WHO CTC.
Number of emergency room visits while using Velcade therapy | Up to 3 years
  Emergency room visits will be considered as a measure of health care resource utilization associated with Velcade therapy.
Number of inpatient hospital stays while using Velcade therapy | Up to 3 years
  Inpatient hospital stays and the reasons for hospitalization will be considered as a measure of health care resource utilization associated with Velcade therapy.
Number of days for each hospital stay | Up to 3 years
  Days for each hospital stay will be considered as a measure of health care resource utilization associated with Velcade therapy.
Number of patients on whom therapeutic therapies will be conducted | Up to 3 years
  Therapeutic therapies (eg: surgery) will be considered as a measure of health care resource utilization associated with Velcade therapy.
Number of patients on whom chest radiograph will be conducted | Up to 3 years
Number of patients on whom whole-body bone scan will be conducted | Up to 3 years
Number of patients on whom radiograph for designated area will be conducted | Up to 3 years
Serum immunoglobin and M-protein | Up to 3 years
M-protein detected by immunofixation electrophoresis | Up to 3 years
Urine light chain M-protein | Up to 3 years
Bone marrow puncture and biopsy | Up to 3 years
β2-microglobulin | Up to 3 years
C-reactive protein | Up to 3 years
Lactate dehydrogenase | Up to 3 years
Routine blood examination | Up to 3 years
Liver function test | Up to 3 years
Renal function test | Up to 3 years
Serum electrolytes | Up to 3 years
Number of patients on concomitant medications | Up to 3 years
  Concomitant medications will be considered as a measure of health care resource utilization associated with Velcade therapy. Concomitant medications include over-the-counter as well as prescription medications, start and stop dates, dosages, and indication. The compliance of concomitant medications will be evaluated by the percentage of patient reported dose over prescribed dose.

SECONDARY OUTCOMES:
Indications for Velcade therapy | Baseline (Day -1)
  Multiple myeloma patients who receive two or more prior treatments and demonstrate disease progression on the most recent treatment will be indicated for Velcade therapy.
Sociodemographics for Velcade therapy | Baseline
  Sociodemographics of patients will be assessed, at the initiation of Velcade therapy, such as: gender, date of birth, height, weight, highest degree, and career information.
Number of chronic concomitant disease | Baseline
  Chronic concomitant disease will be assessed at the initiation of Velcade therapy.
Treatment history | Baseline
  Treatment history will be assessed at the initiation of Velcade therapy. Treatment history includes: confirmation date of diagnosis of multiple myeloma patients or other patients receiving Velcade therapy; names of diseases for patient receiving Velcade therapy; prior treatments for multiple myeloma; outcomes of prior treatments for multiple myeloma.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.

REFERENCES:
- [Derived] Lin M, Hou J, Chen W, Huang X, Liu Z, Zhou Y, Li Y, Zhao T, Wang L, Wu KW, Shen Z. Improved response rates with bortezomib in relapsed or refractory multiple myeloma: an observational study in Chinese patients. Adv Ther. 2014 Oct;31(10):1082-94. doi: 10.1007/s12325-014-0159-z. Epub 2014 Oct 21. PMID 25331616
- See also: VELCADE (Bortezomib for Injection) Observational Study — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1482&filename=CR006373_CSR.pdf